CLINICAL TRIAL: NCT04406506
Title: Comparative Study Between Different Methods of Enteral Feeding in Acute Severe Pancreatitis
Brief Title: Entral Feeding in Acute Severe Pancreatitis
Status: Completed | Type: Observational
Sponsor: King Abdul Aziz Specialist Hospital (Network)
Responsible Party: Sponsor
Other Study IDs: ICU-28-20
Record Dates: First submitted 2020-05-21; First posted 2020-05-28 (Actual); Last update posted 2020-05-28 (Actual); Status verified 2020-05

CONDITIONS: Postoperative Nausea
MeSH Terms: conditions — Postoperative Nausea and Vomiting | interventions — Intubation, Gastrointestinal; Erythromycin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 13 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (2):
- Group A: Group A received nasogastric feeding (NG), insure through ngt pump
  Interventions: Device: nasogastric; Drug: (erythromycin 250 mg IV bolus)
- Group B: * receive feeding throughThe nasojejunal tube is silicone or polyurethane tube with an inner stylet that is positioned (under fluoroscopic guidance) beyond the ligament of Treitz.
  * Patients were placed in right lateral position
  Interventions: Device: nasojejunal; Drug: (erythromycin 250 mg IV bolus)

INTERVENTIONS:
Device: nasogastric — • The insertion of NG tubes were performed by the ICU physician and the position was checked by auscultation of gas from 50 ml syringe by injecting 20 ml of air in the NG and by X-ray abdomen to be sure from the site of NG tube
  Groups: Group A
Device: nasojejunal — * The nasojejunal tube is silicone or polyurethane tube with an inner stylet that is positioned (under fluoroscopic guidance) beyond the ligament of Treitz.
  * Patients were placed in right lateral position
  Groups: Group B
Drug: (erythromycin 250 mg IV bolus) — prokinetic (erythromycin 250 mg IV bolus) given to assist the passage of the tube through the pylorus

SUMMARY:
• A total of 60 patients admitted to King Abdulaziz Specialists Hospital between June 2018 and April 2020 with both a clinical and biochemical presentation of acute pancreatitis with the following inclusion criteria: Abdominal pain > 6 on the visual analogue scale without given analgesia , abdominal distension and tenderness with serum amylase and serum lipase at least 3 times the upper limit of the reference range (considering normal lipase level from 0-160 U/L, and normal amylase level from 0-100 U/L) with confirmed abdominal computerized axial tomography of grade D and E on Ranson and colleagues criteria(28) of inflamed pancreatic picture.

DETAILED DESCRIPTION:
* The study was conducted on monitoring of four pillar for 13 days (data collected one day before feeding and every three days for 12 days). the first pillar comparing the effect of the two enteral feeding methods on the clinical condition of the acute severe pancreatitis and this monitored clinically and laboratory by fixed parameters, clinically, by abdominal pain which assessed by visual analogue scale (VAS). and laboratory, by both markers of severity of pancreatic acini destruction which assessed by serum amylase, lipase and Markers of severity of interstitial pancreatic tissue destruction which assessed by the level of Lactate Dehydrogenase level (LDH), Aspartate aminotransferase (AST), C-reactive protein, prostacyclin and interleukin 8. The second pillar include effect of the two enteral feeding methods on the patient's tolerance and these monitored in our study by both post-feeding vomiting and post feeding attacks of osmotic diarrhea and also abdominal pain. Third pillar include effect of the two enteral feeding methods on the patient's general condition and these monitored by follows the APACHE II Score, hemodynamics of the patients in both groups (Mean arterial blood pressure and pulse) and arterial oxygen saturation (Spo2). Fourth pillar include effect of the two enteral feeding methods on achieving satisfactory nutrition parameters of the patients and both albumin level, radium blood sugar and electrolytes (sodium and potassium level) used as indicator for this.
* All parameters observed one day before starting feeding and every 3 days for 12 days (duration of the study).

ELIGIBILITY:
Inclusion Criteria:

* acute pancreatitis

Exclusion Criteria:

* systemic disease as hypertension or diabetes

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: * A total of 60 patients admitted to King Abdulaziz Specialists Hospital between June 2018 and April 2020 with both a clinical and biochemical presentation of acute pancreatitis with the following inclusion criteria: Abdominal pain > 6 on the visual analogue scale without given analgesia , abdominal distension and tenderness with serum amylase and serum lipase at least 3 times the upper limit of the reference range (considering normal lipase level from 0-160 U/L, and normal amylase level from 0-100 U/L) with confirmed abdominal computerized axial tomography of grade D and E on Ranson and colleagues criteria(28) of inflamed pancreatic picture.
  * An acute physiology and chronic health evaluation (APACHE) II were done for all of them and only score of > 8 included in our study.
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2018-06-10 (Actual); Primary Completion 2020-04-02 (Actual); Study Completion 2020-04-10 (Actual)

PRIMARY OUTCOMES:
effect of different methods of feeding in the clinical condition of the acute severe pancreatitis | 13 days
  first pillar comparing the effect of the two enteral feeding methods on the clinical condition of the acute severe pancreatitis,The second pillar include effect of the two enteral feeding methods on the patient's tolerance

CONTACTS AND LOCATIONS:
Locations (1):
- King abd el Aziz specialist hospital, Ta'if, Saudi Arabia